CLINICAL TRIAL: NCT04591119
Title: Bilateral Transversus Thoracis Muscle Plane Block for Acute Postoperative Pain in Adult Coronary Artery Bypass Graft Surgery: A Randomized Controlled Observer Blinded Trial
Brief Title: Transversus Thoracis Muscle Plane Block for Postoperative Pain in Adult Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Melike Korkmaz Toker, Assistant Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MSKU 20-IV
Record Dates: First submitted 2020-10-11; First posted 2020-10-19 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Pain; Chest Pain; Coronary Artery Bypass; Sternotomy
Keywords: adult cardiac surgery; poststernotomy pain; transversus thoracic muscle plane block; parasternal intercostal block; behavioral pain scale; numeric rating scale
MeSH Terms: conditions — Pain, Postoperative; Chest Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transversus Thoracic Muscle Plane Block (TTMPB) Group (Active Comparator): At the TTMPB group, the block will be performed by the surgeon before the closure of the sternum by visualizing the muscles and identifying them. In the TTMPB group patients will receive 40 ml %0.375 bupivacaine divided into 4 equal doses between internal intercostal muscle and transversus thoracic muscle at the 2nd and 3rd intercostal space and 4th and 5th intercostal space.
  Interventions: Procedure: Transversus Thoracic Muscle Plane Block
- Parasternal Intercostal Block (PSIB) Group (Active Comparator): At the PSIB group, the block will be performed by ultrasound guidance after completion of surgery. PSIB Blocks will be performed under ultrasonography guidance using a linear 6 to 13 megahertz ultrasound probe by the anesthesist.In PSIB group patients will receive 40 ml %0.375 bupivacaine divided into 4 equal doses between psoas major muscle and external intercostal muscle at the 2nd and 3rd intercostal space and 4th and 5th intercostal space bilaterally.
  Interventions: Procedure: Parasternal Intercostal Plane Block
- Control Group (No Intervention): At the control group, no intervention for pain management will be done.

INTERVENTIONS:
Procedure: Transversus Thoracic Muscle Plane Block — 40 ml %0.375 bupivacaine divided into 4 equal doses will be injected by the surgeon between internal intercostal muscle and transversus thoracis muscle at the 2nd and 3rd intercostal space and 4th and 5th intercostal space
  Arms: Transversus Thoracic Muscle Plane Block (TTMPB) Group
Procedure: Parasternal Intercostal Plane Block — 40 ml %0.375 bupivacaine injection will be performed by ultrasound guidance after completion of surgery between pectoralis major muscle and external intercostal muscle at the 2nd and 3rd intercostal space and 4th and 5th intercostal space bilaterally by anesthesiologist.
  Arms: Parasternal Intercostal Block (PSIB) Group

SUMMARY:
Inadequate pain control after coronary artery bypass graft surgery increases mortality and results in a higher incidence of persistent poststernotomy pain syndrome. Our aim is to assess whether ultrasound-guided parasternal intercostal block (PSIB) or surgeon implied transversus thoracic muscle plane block (TTMPB) would improve the postoperative pain scores and decrease tramadol consumption better after coronary artery bypass graft surgery

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status II-III
* Elective coronary artery bypass graft surgery under general anesthesia

Exclusion Criteria:

* American Society of Anesthesiologists physical status IV
* Emergency surgery and redo surgery
* Low cardiac output syndrome, perioperative intra-aortic balloon pump support for any reason, bleeding disorder or abnormal coagulation profile, abnormal hepatic and renal parameters, uncontrolled diabetes mellitus, chronic obstructive pulmonary disease, atrial fibrillation on anticoagulation
* Allergy to any study drugs, local infection at the block site
* Opioid abuse

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | Postoperative 24th hour
  Tramadol consumption will be assessed by checking patient daily drug order records
Postoperative opioid consumption | Postoperative 1st, 4th and 12th hour
  Tramadol consumption will be assessed by checking patient daily drug order records

SECONDARY OUTCOMES:
Behavioral Pain Scale | postoperative 1st and 4th hour
  A blinded nurse will assess postoperative pain while they are intubated at the 1st and 4th hour by using 3 subscale Behavioral Pain Scale which ranges from 3 (no pain) to 12 (maximum pain)
Numeric Rating Scale | Postoperative 12th and 24th hour
  A blinded nurse will assess postoperative pain during resting and movement at postoperative 12th and 24th hour by using Numeric rating scale at the extubated patient by using 11-point Numerical Rating Scale which ranges from '0' (means no pain) to '10' (means worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Melike Korkmaz Toker, Assist.Prof, Principal Investigator — Mugla Sıtkı Kocman University Department of Anesthesiology and Reanimation
Locations (1):
- Mugla Sıtkı Kocman University Training nad research Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
via mail

REFERENCES:
- [Background] Ueshima H, Takeda Y, Ishikawa S, Otake H. RETRACTED: Ultrasound-guided transversus thoracic muscle plane block: a cadaveric study of the spread of injectate. J Clin Anesth. 2015 Dec;27(8):696. doi: 10.1016/j.jclinane.2015.05.013. Epub 2015 Jul 3. No abstract available. PMID 26144912 (Retraction: PMID 35396105 J Clin Anesth. 2022 Aug;79:110781)
- [Background] de la Torre PA, Garcia PD, Alvarez SL, Miguel FJ, Perez MF. A novel ultrasound-guided block: a promising alternative for breast analgesia. Aesthet Surg J. 2014 Jan 1;34(1):198-200. doi: 10.1177/1090820X13515902. No abstract available. PMID 24396082